CLINICAL TRIAL: NCT06275347
Title: Comparative Study of the Response to Weight Loss and Metabolic Conditions Using Two Non-pharmacological Nutritional Programs
Brief Title: Very Low Calorie Ketogenic Low-fat Diet (VLCKLFD)
Acronym: Zelé2021
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Veracruzana (Other)
Responsible Party: Principal Investigator, Francisco J. Nachón García, MD. PhD Senior Researcher of the Institute of Health Sciences at Universidad Veracruzana Xalapa, Universidad Veracruzana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19CI 30 087 041; 1/1142021 (Other: Comite del Centro de alta especialidad del Estado de Veracruz)
Record Dates: First submitted 2023-12-08; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: A Randomized Clinical Trial was conducted in patients with obesity type I patients
Who Masked: Participant, Care Provider
Masking Description: Eligible patients were assigned to a one of the four VIME Weight Loss and Wellness Center for management and follow up according to their preference, a sequential number in inclusion order was given, with all the patients coded with a 4-digit number. This code was sent to the people in the food production plant where the patients were randomized in a double blinded study, with a 2:1 allocation for low-fat, normo-protein, controlled ketogenic diet (Zélé method) or low calories diet
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Very low calorie ketogenic low-fat diet (VLCKLFD) (Experimental): Frank ketosis: between 650 and 730 kcal/day in 5 mealtimes. This stage in the nutritional intervention was done during the first 4 weeks.
  Mixed Ketosis: in this stage, one intake of commercial preparations was replaced by proteins, which discreetly increased by 100 to 150 Kcal/day. This stage was done during the next 4 weeks.
  Interventions: Other: Low-fat normoprotein Controlled Ketogenic Diet.
- Low-Calorie Diet (LCD) (Active Comparator): The usual caloric intake of a balanced LCD is between 1,200 and 1,500 kcal per day with a macronutrient distribution of 50% carbohydrates, 25% proteins and 25% fats, according to the Diogenes study
  Interventions: Other: Hypocaloric Balanced Diet

INTERVENTIONS:
Other: Low-fat normoprotein Controlled Ketogenic Diet. — Frank ketosis will consist of between 650 and 730 kcal/day in 5 meal times, based on commercial and vegetable preparations with low glycemic index, an average of 1.2 g of protein/kg of ideal weight/day, 20 g/day of lipids based on essential fatty acids and less than 60 g/day of absorbable carbohydrates. Patients will receive vitamin and sodium chloride, magnesium oxide, calcium carbonate. Mixed Ketosis one or two intakes of commercial preparations will be progressively replaced by proteins, which will increase by 100 to 150 Kcal/day, supplementation of vitamins and minerals will continue. Transition Stage simple carbohydrates and some complex carbohydrates are added to the previous program, in an approximate proportion of 30 to 35% protein, 25% fat and 40 to 45 % carbohydrates. Integral and maintenance phase: may vary between 1300 and 2250 kcal/day, with a macronutrient distribution of 50% carbohydrates, 25% proteins and 25% fats.
  Other Names: Zelé
  Arms: Intervention Very low calorie ketogenic low-fat diet (VLCKLFD)
Other: Hypocaloric Balanced Diet — Balanced hypocaloric diet (caloric intake 20% below basal metabolic expenditure measured by Multifrequency Bioelectrical Impedance or calculated according to the FAO/WHO/UN formula (FAO/WHO/UNU (1985). Energy and Protein requirements. Technical Report Series No 724, World Health Organization, Geneva). The usual caloric intake of a balanced hypocaloric diet is between 1,200 and 1,400 kcal per day with a macronutrient distribution of 50% carbohydrates, 25% proteins and 25% fats, according to the Diogenes study
  Other Names: Low-Calorie Diet (CD)
  Arms: Low-Calorie Diet (LCD)

SUMMARY:
This study aimed to assess the efficacy and safety of the Zélé program, a controlled ketogenic diet, for weight loss and maintenance. It involved a randomized clinical trial with participants aged 18-60, BMI between 30-34.9 kg/m², and no severe health issues

DETAILED DESCRIPTION:
The study will be conducted in Mexico City under the sponsorship of Zélé® and in collaboration with the VIME Weight Loss and Wellness Center of Mexico. During the year 2021 and with follow-up for 24 months. An open call will be made through different media including social networks for the recruitment of patients who meet the inclusion criteria and must present themselves for a clinical evaluation in which pathological history, clinical status, heart rate, blood pressure, oxygenation and temperature will be recorded. Nutritional assessment, and a Complete Blood Count, a biochemical profile. Patients who meet all the inclusion criteria will be selected and will have an interview with the principal investigator in which they will sign their letter of commitment and informed consent, then they will be subjected to the randomization process with a 2:1 allocation for treatment and controls, respectively. Subsequently, they will be submitted to the two nutritional treatments and will be clinically evaluated every week and will receive nutritional, psycho emotional and physical activity counseling. At each visit, adverse effects, changes in clinical status will be recorded and the presence of ketone bodies in capillary blood will be determined. Subsequently, only clinical and nutritional follow-up will be given along with psycho-emotional support and physical activity advice every 3 months up to 12 months and every 6 months up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex, between 18 and 60 years old, with a body mass index (BMI) between 30 and 34.9 kg/m2 were eligible to participate in the study. We recruited participants from Mexico City through different media including social networks (Facebook and Instagram). The selection was consecutive according to the order of response of the interested participants. All participants read and signed the Informed Consent form

Exclusion Criteria:

* Pregnant or breastfeeding patients, patients with severe eating disorders, alcoholism, or drug addiction, patients with severe psychiatric disorders (e.g., schizophrenia, bipolar disorder, mayor depression), patients with hepatic alteration defined as increase of ALT, AST, GGT more than 4 folds the reference value, patients with renal impairment defined as a glomerular filtration rate below 60 ml/min. Patients with type 1 or insulin-dependent DM, or DM2 on insulin therapy, patients with obesity caused by endocrinological diseases (except type 2 DM), patients with hemopathies, cancer patients, patients with active cardiovascular or cerebrovascular disease (heart rhythm disorders, recent infarction [<6m], unstable angina, decompensated heart failure, recent vascular accident [<6m]), patients with gout, patients with known renal lithiasis or cholelithiasis, patients with electrolyte disorders, patients with orthostatic hypotension, patients with known an altered or abnormal electrocardiogram.

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of this nutritional intervention | Every week for 4 months, then every month for two years
  The primary outcome measure was body weight operationalized as the change in an individual's mass or weight loss in kilograms.
Volume of total body tissue corresponding to muscle | Every week for 4 months, then every month for two years
  It will be measured with unit Kilogram, minimun 10, maximum 150, with a Multi-frequency Bioelectrical Impedance Equipment
Percentage of body weight made up of adipose tissue | Every week for 4 months, then every month for two years
  It will be measured with unit percentaje, minimum 9, maximum 90, with a Multi-frequency Bioelectrical Impedance Equipment
Visceral Fat | Every week for 4 months, then every month for two years
  It will be measured with unit index, from 1 to 40, with a Multi-frequency Bioelectrical Impedance Equipment
Bone mass | Every week for 4 months, then every month for two years
  the skeletal weight will be measured with unit kilograms (kg), from 1 to 70 kg, with a Multi-frequency Bioelectrical Impedance Equipment
Total body water | Every week for 4 months, then every month for two years
  Percentage of the body that corresponds to water, unit % (percentaje) and/ or kilograms (kg) from 0 to 150 with a Multi-frequency bioelectrical impedance equipment
Waist circumference | Every week for 4 months, then every month for two years
  Measurement made with a tape measure directly on the skin (without clothing). It will be measured at the height of the middle of the armpit, at the point between the bottom of the last rib and the highest part of the hip. Unit centimeters (cm), minimum 30, maximum 200, Using tape measure
Hip circumference | Every week for 4 months, then every month for two years
  Circumference of the widest part above the buttocks. Unit cm, minimum 30, maximum 200. Measuring with tape measure
Muscular strenght | Every week for 4 months, then every month for two years
  Isometric muscle strenght in the dominant hand, unit kilograms (kg)/ Strength, registration form digital dynamometer
Weight | Every week for 4 months, then every month for two years
  it will be measured in unit kilograms, in a weighing machine
Height | Every week for 4 months, then every month for two years
  The size will be measured in meters with a stadiometer
BMI Body index mass | Every week for 4 months, then every month for two years
  Body mass index is an index composed of weight/height squared in kg/m2.

SECONDARY OUTCOMES:
Hemoglobin | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a Clinical laboratory determination, unit gr/L (grams/liters)
Hematocrit | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a Clinical laboratory determination, unit percentage (%), minimumm 10, maximum 16
Leukocytes | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a Clinical laboratory determination, unit quantity per cc, minimumm 4000, maximum 18000.
Fasting Blood Glucose | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mg/dl (miligrams/deciliters), Normoglycemia in fasting 70 to 100 mg/dl. Hyperglycemia higher than 100 mg/dl in fasting. Diabetes 126 mg/Dl of fasting blood glucose.
Glycated hemoglobin (HbA1c) | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit percentage (%), 6% very low, 7% moderate, 8% high, 9% very high, 10% risk.
Insulin | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit UI/ml (Interantional unit/ mililiter), hyperinsulinemia >6UI/ml
Creatinine | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mg/dl (miligrams/deciliters), minimum 0.4, maximum 1.3
Urea | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mg/dl (miligrams/deciliters), minimum 8, maximum 54
Uric acid | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mg/dl (miligrams/deciliters), minimum 2.4, maximum 9.
Sodium | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mEq/l (miliequivalents/ litre), minimum 90, maximum 110.
Potassium | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mEq/l (miliequivalents/ litre), minimum 3.5, maximum 5.5
Calcium | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mg/dl (miligrams/ deciliters), minimum 8.5, maximum 10.5
Phosphorus | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mg/dl (miligrams/ deciliters), minimum 2.5, maximum 4.5,
Magnesium | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mg/dl (miligrams/ deciliters), minimum 1.5, maximum 2.5,
Albumin | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mg/dl (miligrams/ deciliters), minimum 3.4, maximum 5.4,
Direct bilirubin | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mg/dl (miligrams/ deciliters), normal value less than 0.3 mg/dl (0 less than 5.1mg/dl)
Indirect bilirubin | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mg/dl (miligrams/ deciliters), minimum 0.1, maximum 0.5
Total bilirubin | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mg/dl (miligrams/ deciliters), minimum 0.1, maximum 1.2
Alanine aminotransferase | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit IU/L (interantional unit/ liters), minimum 10, maximum 41.
Aspartate Amino Transferase | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit IU/L (interantional unit/ liters), minimum 5, maximum 37
Total cholesterol | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mg/dl (miligrams/ deciliters), minimum 100, maximum 200
Triglycerides | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mg/dl (miligrams/ deciliters), minimum 100, maximum 500
High Density Lipoproteins | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mg/dl (miligrams/ deciliters), greater than 40 mg/dl
Low Density lipoproteins | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mg/dl (miligrams/ deciliters), less than 100 mg/dl
Protein C Reactive | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mg/dl (miligrams/ deciliters), less than 10 mg/dl
Thyroid stimulating hormone | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit IU/L (interantional unit/ liters), from 0.3 to 3 IU
Triiodothyronine | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit IU/L (nanograms/ mililiters), from 0.8 to 2 ng/ml
Thyroxine | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit pg/ml (picograms/ mililiters), from 5.4 to 11.5 pg/ml
Cholecalciferol | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit ng/ml (nanograms/ mililiters), from 25 to 90 ng/ml
Gasometric variables, Partial pressure of oxygen (PaO2) | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mmHg (milimeters of mercury), minimum 75, maximum 100
HCO3 (Bicarbonate ion plasma concentration) | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mEq/L (miliequivalents per litre), minimum 21, maximum 30
Arterial pH | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, minimum 7.35, maximum 7.45
Lactic acid | Every 2 months for the first 6 months, then every 6 months for two years
  It will be measured by a blood tests, unit mg/L (miligrams/liters), from 4.5 to 19 mg/L

OTHER OUTCOMES:
Adherence to this nutritional intervention | Every week for 4 months, then every month for a two years
  It will be measured by complied or did not comply with the program, making a question.
Satisfaction survey | Every week for 4 months, then every month for a two years
  Interrogation very satified to very dissatisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Francisco J Nachón García, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palgi A, Read JL, Greenberg I, Hoefer MA, Bistrian BR, Blackburn GL. Multidisciplinary treatment of obesity with a protein-sparing modified fast: results in 668 outpatients. Am J Public Health. 1985 Oct;75(10):1190-4. doi: 10.2105/ajph.75.10.1190. PMID 4037162
- [Background] Hemmingsson E, Johansson K, Eriksson J, Sundstrom J, Neovius M, Marcus C. Weight loss and dropout during a commercial weight-loss program including a very-low-calorie diet, a low-calorie diet, or restricted normal food: observational cohort study. Am J Clin Nutr. 2012 Nov;96(5):953-61. doi: 10.3945/ajcn.112.038265. Epub 2012 Sep 18. PMID 22990030
- [Background] Lartey S, Si L, Lung T, Magnussen CG, Boateng GO, Minicuci N, Kowal P, Hayes A, de Graaff B, Blizzard L, Palmer AJ. Impact of overweight and obesity on life expectancy, quality-adjusted life years and lifetime costs in the adult population of Ghana. BMJ Glob Health. 2020 Sep;5(9):e003332. doi: 10.1136/bmjgh-2020-003332. PMID 32994229
- [Background] Foster D, Sanchez-Collins S, Cheskin LJ. Multidisciplinary Team-Based Obesity Treatment in Patients With Diabetes: Current Practices and the State of the Science. Diabetes Spectr. 2017 Nov;30(4):244-249. doi: 10.2337/ds17-0045. PMID 29151714
- [Result] Pirozzo S, Summerbell C, Cameron C, Glasziou P. Should we recommend low-fat diets for obesity? Obes Rev. 2003 May;4(2):83-90. doi: 10.1046/j.1467-789x.2003.00099.x. PMID 12760443
- [Result] Blackburn GL, Bistrian BR. Careers in nutrition from the clinical viewpoint. Nutr Rev. 1976 Apr;34(4):97-104. doi: 10.1111/j.1753-4887.1976.tb05719.x. No abstract available. PMID 817237
- [Result] Tsai AG, Wadden TA. The evolution of very-low-calorie diets: an update and meta-analysis. Obesity (Silver Spring). 2006 Aug;14(8):1283-93. doi: 10.1038/oby.2006.146. PMID 16988070
- [Result] Goday A, Bellido D, Sajoux I, Crujeiras AB, Burguera B, Garcia-Luna PP, Oleaga A, Moreno B, Casanueva FF. Short-term safety, tolerability and efficacy of a very low-calorie-ketogenic diet interventional weight loss program versus hypocaloric diet in patients with type 2 diabetes mellitus. Nutr Diabetes. 2016 Sep 19;6(9):e230. doi: 10.1038/nutd.2016.36. PMID 27643725
- [Result] Elfhag K, Rossner S. Initial weight loss is the best predictor for success in obesity treatment and sociodemographic liabilities increase risk for drop-out. Patient Educ Couns. 2010 Jun;79(3):361-6. doi: 10.1016/j.pec.2010.02.006. Epub 2010 Mar 11. PMID 20223613
- [Result] Handjieva-Darlenska T, Handjiev S, Larsen TM, van Baak MA, Jebb S, Papadaki A, Pfeiffer AF, Martinez JA, Kunesova M, Holst C, Saris WH, Astrup A. Initial weight loss on an 800-kcal diet as a predictor of weight loss success after 8 weeks: the Diogenes study. Eur J Clin Nutr. 2010 Sep;64(9):994-9. doi: 10.1038/ejcn.2010.110. Epub 2010 Jun 30. PMID 20588292
- [Result] Nackers LM, Ross KM, Perri MG. The association between rate of initial weight loss and long-term success in obesity treatment: does slow and steady win the race? Int J Behav Med. 2010 Sep;17(3):161-7. doi: 10.1007/s12529-010-9092-y. PMID 20443094
- [Result] Blackburn GL. Weight of the nation: moving forward, reversing the trend using medical care. Am J Clin Nutr. 2012 Nov;96(5):949-50. doi: 10.3945/ajcn.112.049643. Epub 2012 Oct 3. No abstract available. PMID 23034956
- [Result] Larsen TM, Dalskov SM, van Baak M, Jebb SA, Papadaki A, Pfeiffer AF, Martinez JA, Handjieva-Darlenska T, Kunesova M, Pihlsgard M, Stender S, Holst C, Saris WH, Astrup A; Diet, Obesity, and Genes (Diogenes) Project. Diets with high or low protein content and glycemic index for weight-loss maintenance. N Engl J Med. 2010 Nov 25;363(22):2102-13. doi: 10.1056/NEJMoa1007137. PMID 21105792
- [Result] Cano-Rodríguez I, Ballesteros-Pomar MD, Pérez-Corral B, Aguado R. Dietas bajas en hidratos de carbono frente a dietas bajas en grasas. Endocrinol Nutr 2006;53(3):209-17 dol: http://dx.doi.org/10.1016/s1575-0922(06)71091-9
- [Result] Joint WHO/FAO/UNU Expert Consultation. Protein and amino acid requirements in human nutrition. World Health Organ Tech Rep Ser. 2007;(935):1-265, back cover. PMID 18330140
- [Result] Díaz-Muñoz GA, Castañeda-Gómez ÁM, Belalcázar-Monsalve MP, Zambrano-Salazar JP, Bautista-Velandia MC, Ballesteros-Arbeláez F. Efecto de la dieta cetogénica baja en calorías sobre la composición corporal en adultos con sobrepeso y obesidad: revisión sistemática y metaanálisis. Rev Nutr Clin Metab. 2021;4(3):98-113. http://dx.doi.org/10.35454/rncm.v4n3.273
- [Result] Merra G, Gratteri S, De Lorenzo A, Barrucco S, Perrone MA, Avolio E, Bernardini S, Marchetti M, Di Renzo L. Effects of very-low-calorie diet on body composition, metabolic state, and genes expression: a randomized double-blind placebo-controlled trial. Eur Rev Med Pharmacol Sci. 2017 Jan;21(2):329-345. PMID 28165552
- [Result] Romano L, Marchetti M, Gualtieri P, Di Renzo L, Belcastro M, De Santis GL, Perrone MA, De Lorenzo A. Effects of a Personalized VLCKD on Body Composition and Resting Energy Expenditure in the Reversal of Diabetes to Prevent Complications. Nutrients. 2019 Jul 4;11(7):1526. doi: 10.3390/nu11071526. PMID 31277506
- [Result] Colombo O, Ferretti VV, Ferraris C, Trentani C, Vinai P, Villani S, Tagliabue A. Is drop-out from obesity treatment a predictable and preventable event? Nutr J. 2014 Feb 3;13:13. doi: 10.1186/1475-2891-13-13. PMID 24490952
- [Result] Moreno B, Crujeiras AB, Bellido D, Sajoux I, Casanueva FF. Obesity treatment by very low-calorie-ketogenic diet at two years: reduction in visceral fat and on the burden of disease. Endocrine. 2016 Dec;54(3):681-690. doi: 10.1007/s12020-016-1050-2. Epub 2016 Sep 13. PMID 27623967
- [Result] Sajoux I, Lorenzo PM, Gomez-Arbelaez D, Zulet MA, Abete I, Castro AI, Baltar J, Portillo MP, Tinahones FJ, Martinez JA, Crujeiras AB, Casanueva FF. Effect of a Very-Low-Calorie Ketogenic Diet on Circulating Myokine Levels Compared with the Effect of Bariatric Surgery or a Low-Calorie Diet in Patients with Obesity. Nutrients. 2019 Oct 4;11(10):2368. doi: 10.3390/nu11102368. PMID 31590286
- See also: Short-term safety, tolerability and efficacy of a very low-calorie-ketogenic diet interventional weight loss program versus hypocaloric diet in patients with type 2 diabetes mellitus. — http://dx.doi.org/10.1038/nutd.2016.36
- See also: Initial weight loss is the best predictor for success in obesity treatment and sociodemographic liabilities increase risk for drop-out — http://dx.doi.org/10.1016/j.pec.2010.02.006
- See also: Initial weight loss on an 800-kcal diet as a predictor of weight loss success after 8 weeks: the Diogenes study. — http://dx.doi.org/10.1038/ejcn.2010.110
- See also: The association between rate of initial weight loss and long-term success in obesity treatment: Does slow and steady win the race? — http://dx.doi.org/10.1007/s12529-010-9092-y
- See also: Weight of the nation: moving forward, reversing the trend using medical care — http://dx.doi.org/10.3945/ajcn.112.049643
- See also: Dietas bajas en hidratos de carbono frente a dietas bajas en grasas. — http://dx.doi.org/10.1016/s1575-0922(06)71091-9
- See also: Efecto de la dieta cetogénica baja en calorías sobre la composición corporal en adultos con sobrepeso y obesidad: revisión sistemática y metaanálisis — http://dx.doi.org/10.35454/rncm.v4n3.273

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT06275347/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT06275347/ICF_001.pdf